CLINICAL TRIAL: NCT00291473
Title: Safety and Immunogenicity of Cholesterol-Bearing Hydrophobized Pullulan HER2 Protein 146 (CHP-HER2) and NY-ESO-1 Protein (CHP-NY-ESO-1) in Combination With OK-432 in HER2- and/or NY-ESO-1-Expressing Cancers
Brief Title: Safety and Immunogenicity of CHP-HER2 and CHP-NY-ESO-1 Protein With OK-432 in Antigen-Expressing Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Mie University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LMT2004-011
Record Dates: First submitted 2006-02-10; First posted 2006-02-14 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-03

CONDITIONS: Esophageal Cancer; Lung Cancer; Stomach Cancer; Breast Cancer; Ovarian Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Lung Neoplasms; Stomach Neoplasms; Breast Neoplasms; Ovarian Neoplasms

INTERVENTIONS:
Drug: CHP-HER2, CHP-NY-ESO-1

SUMMARY:
Mixed cancer vaccines, CHP-HER2 protein and CHP-NY-ESO-1 protein, are to be studied to evaluate the safety and immune responses in patients who are positive either or both antigens. Nine patients will be enrolled, who are refractory to standard therapies for cancer or at high risk to relapse. CHP-HER2 and CHP-NY-ESO-1 are subcutaneously given on bimonthly basis, together with OK-432(Picibanil) as an immunoadjuvant. Six doses will be given. Toxicity profiles will be monitored, and antigen specific humoral anad T cell responses will be described.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of cancer.
2. HER2 expression in tumor cells scored as 1+ or more which should be confirmed by IHC using at least two antibodies (archived issue; see Appendix 1 and Reference 1 for methodology).

   or NY-ESO-1 expression by reverse transcriptase and polymerase chain reaction (RT-PCR) analysis (Appendix 2), preferably, or immunohistochemistry
3. Patients must

   1. are at high risk of recurrence, more than 25% of probability, after complete resection or even after post-operative adjuvant treatment, and effective adjuvant therapy is not available or refused; or
   2. have metastatic disease, and treatment has failed, or in the situation where effective therapy is not available, or has been refused.
4. Complete recovery from surgery (at least 4 weeks).
5. Laboratory values within the following limits:

   Hemoglobin 9.0 g/dL or more, or 10.0 g/dL or more if <50 kg Neutrophil count >1.5 x 109/L Lymphocyte count >0.5 x 109/L Platelet count >100 x 109/L Serum creatinine ≤ 1.8 mg/dL Serum bilirubin ≤ 2 mg/dL
6. Performance status > 70 (Karnofsky Scale) and life expectancy >3 months.
7. Age 18 years or more.

Exclusion Criteria:

1. Clinically significant heart disease (NYHA Class III or IV).
2. Cardiac dysfunction; less than 50% of ejection fraction by echocardiogram.
3. Immunodeficiency disease.
4. Other serious illnesses, eg, serious infections requiring antibiotics, bleeding disorders.
5. Previous bone marrow or stem cell transplant.
6. Metastatic disease to the central nervous system, unless treated and stable.
7. known HIV antibody positivity.
8. Anaphylactic reaction to previous vaccination.
9. Hypersensitivity to penicillin
10. Chemotherapy, any type of radiation therapy, or immunotherapy within 4 weeks before study entry (6 weeks for nitrosoureas).
11. Concomitant treatment with steroids. Topical or inhalational steroids are permitted.
12. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.
13. Pregnancy or nursing .
14. Refusal, by women of childbearing potential, to use medically acceptable means of contraception.
15. Mental impairment that may compromise the ability to give informed consent.
16. Lack of availability for immunological and clinical follow-up assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2005-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
adverse events

SECONDARY OUTCOMES:
immune responses including HER2 and NY-ESO-1 specific IgG and T cells

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Shiku, M.D., Principal Investigator — Mie University
Locations (1):
- Mie University Hospital, Tsu, Mie-ken, Japan